CLINICAL TRIAL: NCT00503724
Title: Phase I and Pharmacokinetic Study of Enzastaurin (LY317615) in Children and Adolescents With Refractory Primary CNS Tumors
Brief Title: Enzastaurin in Treating Young Patients With Refractory Primary CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000557572; U01CA081457 (NIH); PBTC-023 (Other: Pediatric Brain Tumor Consortium)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma
Keywords: recurrent childhood brain stem glioma; childhood central nervous system germ cell tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; childhood oligodendroglioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood pineoblastoma; recurrent childhood brain tumor; disseminated neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Medulloblastoma; Oligodendroglioma; Optic Nerve Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: enzastaurin hydrochloride — Participants receive 200, 260, 340, or 440 mg/m2/day of enzastaurin orally once daily for 28 days (one course) during the dose escalation phase of the study. To study the toxicity profile of the MTD or phase II recommended dose established during the dose escalation phase, participants receive twice daily doses of enzastaurin orally at the phase II recommended dose for 28 days (one course). In the absence of unacceptable toxicity or disease progression, treatment may continue for 13 courses (approximately one year).
  Other Names: LY317615 monohydrochloride

SUMMARY:
RATIONALE: Enzastaurin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of enzastaurin in treating young patients with refractory primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum tolerated dose (MTD) and/or recommend a phase II dose of enzastaurin hydrochloride in children with recurrent or refractory CNS tumors who are not receiving enzyme-inducing anticonvulsants.
* To further characterize the pharmacokinetics and toxicity of the recommended phase II dose of enzastaurin hydrochloride given twice daily in these patients.

Secondary

* To characterize the pharmacokinetics of enzastaurin hydrochloride at the recommended phase II dose given once a day or twice a day in children.
* To document and describe toxicities associated with enzastaurin hydrochloride.
* To document antitumor activity in children with recurrent or refractory CNS tumors.
* To explore changes in MR perfusion scans obtained within 15 ± 2 days after initiation of enzastaurin hydrochloride therapy as compared to baseline and to correlate these changes with clinical outcome.
* To evaluate a panel of biological surrogate markers in this patient population at baseline and following enzastaurin hydrochloride administration.

OUTLINE: This is a multicenter study.

Patients receive oral enzastaurin hydrochloride once daily until the maximum tolerated dose (MTD) is determined. Patients then receive enzastaurin hydrochloride at the MTD twice daily on days 1-28. Treatment repeats every 28 days for 13 courses in the absence of disease progression or unacceptable toxicity. Patients may receive 13 additional courses (for a total of 26 courses) of oral enzastaurin hydrochloride if the patient is benefitting from the treatment and the investigator and subject agree to continue treatment.

Patients undergo blood sample collection periodically for pharmacokinetic studies.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS malignancy including low-grade glioma

  * All tumors, except intrinsic brain stem and diffuse optic pathway tumors, must have histological verification at either the time of diagnosis or recurrence

    * Patients with intrinsic brain stem or diffuse optic pathway tumors must have clinical and/or radiographic evidence of progression
* Recurrent or progressive disease or disease refractory to standard therapy and for which there is no known curative therapy

PATIENT CHARACTERISTICS:

Inclusion Criteria:

* Karnofsky performance scale (for > 16 years of age) or Lansky performance score (for ≤ 16 years of age) ≥ 60% assessed within two weeks prior to registration
* Peripheral absolute neutrophil count (ANC) ≥ 1,000/μL
* Platelet count ≥ 100,000/μL (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR maximum serum creatinine based on age as follows:

  * 0.8 mg/dL (≤ 5 years of age)
  * 1.0 mg/dL (6 to 10 years of age)
  * 1.2 mg/dL (11 to 15 years of age)
  * 1.5 mg/dL (≥ 16 years of age)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* ALT ≤ 5 x ULN for age
* Serum albumin ≥ 2.5 g/dL
* Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Negative pregnancy test
* Patients must have a normal QTc for age and no evidence of a clinically significant arrhythmia on ECG
* No evidence of active graft-versus-host disease

Exclusion Criteria:

* Pregnant or lactating
* Body surface area < 0.5 m^2
* Clinically significant unrelated systemic illness that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results
* Known hypersensitivity to enzastaurin hydrochloride or its components
* Inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy

PRIOR CONCURRENT THERAPY:

Inclusion Criteria:

* Must have recovered from the acute toxic effects (grade ≤ 2) of all prior therapy before entering this study
* Must not have received myelosuppressive chemotherapy within 3 weeks of entry onto this study (6 weeks for prior nitrosourea)
* At least 7 days since the completion of therapy with a hematopoietic growth agent (i.e., filgrastim [G-CSF], sargramostim [GM-CSF], or erythropoietin)

  * At least 14 days since long-acting formulations
  * Therapeutic use of myeloid growth factors in patients with serious neutropenic conditions, such as sepsis, may be considered at the investigator's discretion
* At least 7 days since the completion of therapy with a biologic agent
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months must have elapsed after prior total body irradiation (TBI) or craniospinal radiotherapy
* At least 6 weeks must have elapsed after other substantial bone marrow irradiation
* At least 6 months since prior allogeneic bone marrow transplantation
* At least 3 months since prior autologous bone marrow or stem cell transplantation
* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration

  * Corticosteroids should be used at the lowest dose to control symptoms of edema and mass effect

Exclusion Criteria:

* Routine concurrent use of growth factors (i.e., G-CSF, GM-CSF, or erythropoietin)
* Any other concurrent anticancer or investigational drug therapy
* Concurrent enzyme-inducing anticonvulsants (EIACDs)
* Concurrent gents that prolong the QTc
* Concurrent drugs that are substrates or inhibitors of CYP3A4 or CYP2C9
* Other concurrent drugs that are sensitive substrates of CYP2C8, CYP2C9, or CYP2C19 and/or have a narrow therapeutic window

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | First 28 days of therapy
  The maximum tolerated dose or recommended phase II dose will be based on the dose-limiting toxicities observed during the first 28 days of therapy in those participants receiving enzastaurin on a once per day dosing schedule.
Number of participants treated with the maximum tolerated dose or phase II recommended dose on a twice daily dosage schedule with dose-limiting toxicities | First 28 days of therapy

SECONDARY OUTCOMES:
Pharmacokinetics | Three days prior to course 1 and day 28 of course 1
  Blood samples for pharmacokinetic studies will be drawn 3 days prior to course 1 and on day 28 of course 1.
Toxicity | From day 1 of therapy until 30 days after the last dose of the drug
Tumor response | Pre-treatment, day 15 of course 1, and at the end of courses 3, 5, 8, 11, and 13.
  Brain images to assess tumor response (complete response, partial response, or stable disease) are taken pre-treatment, at day 15 of course 1, and at the end of courses 3, 5, 8, 11, and 13.
Change in MR perfusion parameters obtained within 15 ± 2 days after initiation of enzastaurin hydrochloride therapy as compared to baseline | Baseline and day 15 of course 1
Change from baseline in the inhibition of Akt cell signaling at day 14 and day 28 | Pre-treatment and at days 14 and 28 of course 1
Akt pathway activity in pre-study tumor samples | Pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Blaney, MD, Study Chair — Texas Children's Cancer Center
Locations (8):
- United States (8):
  - UCSF Medical Center at Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas